CLINICAL TRIAL: NCT01088711
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK3102 in Obese Subjects and in Patients With Type 2 Diabetes
Brief Title: Evaluation of Omarigliptin (MK-3102) in Obese Participants and in Participants With Type 2 Diabetes (MK-3102-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3102-004
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes (T2D)
Keywords: Type 2 diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Omarigliptin (Experimental): Obese healthy participants receive once-weekly omarigliptin 50 mg by mouth for 4 weeks (Panel A).
  Interventions: Drug: Omarigliptin
- Healthy Placebo (Placebo Comparator): Obese healthy participants receive once-weekly placebo by mouth for 4 weeks (Panel A).
  Interventions: Drug: Placebo
- T2D Omarigliptin (Experimental): Obese participants with T2D receive once-weekly omarigliptin 50 mg by mouth for 4 weeks (Panel B).
  Interventions: Drug: Omarigliptin
- T2D Placebo (Placebo Comparator): Obese participants with T2D receive once-weekly placebo by mouth for 4 weeks (Panel B).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omarigliptin — Once-weekly 50 mg capsule
  Other Names: MK-3102
  Arms: Healthy Omarigliptin; T2D Omarigliptin
Drug: Placebo — Once-weekly placebo capsule
  Arms: Healthy Placebo; T2D Placebo

SUMMARY:
This study will test the safety and tolerability of omarigliptin. It is hypothesized that administration of once-weekly omarigliptin in obese but otherwise healthy participants, and in obese participants with Type 2 diabetes (T2D) will be sufficiently safe and well tolerated to permit continued clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* obese (body mass index [BMI] ≥30 kg/m² and ≤40 kg/m²) male participants and female participants of non-childbearing potential
* has been diagnosed with T2D (Panel B)
* is not actively participating in a weight loss program

Exclusion Criteria:

* has a history of clinically-significant disease (other than T2D)
* has a history of cancer
* has estimated creatinine clearance ≤60 mL/min
* is unable to refrain from or anticipates the use of any prescription or non-prescription medication
* consumes excessive amounts of alcohol or caffeine
* has participated in a previous omarigliptin study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03-11 (Actual); Primary Completion 2010-05-11 (Actual); Study Completion 2010-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Addy C, Tatosian D, Glasgow XS, Gendrano IN 3rd, Kauh E, Martucci A, Johnson-Levonas AO, Selverian D, Matthews CZ, Gutierrez M, Wagner JA, Aubrey Stoch S. Pharmacokinetic and Pharmacodynamic Effects of Multiple-dose Administration of Omarigliptin, a Once-weekly Dipeptidyl Peptidase-4 Inhibitor, in Obese Participants With and Without Type 2 Diabetes Mellitus. Clin Ther. 2016 Mar;38(3):516-30. doi: 10.1016/j.clinthera.2015.12.020. Epub 2016 Feb 9. PMID 26869191
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3102-004&kw=3102-004&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants - Omarigliptin: Obese healthy participants received once-weekly omarigliptin for 4 weeks.
- Healthy - Placebo: Obese healthy participants received once-weekly placebo for 4 weeks.
- T2D - Omarigliptin: Obese T2D participants received once-weekly omarigliptin for 4 weeks.
- T2D - Placebo: Obese T2D participants received once-weekly placebo for 4 weeks.
Period: Overall Study
Arm/Group | Healthy Participants - Omarigliptin | Healthy - Placebo | T2D - Omarigliptin | T2D - Placebo
Started | 18 | 6 | 6 | 2
Completed | 18 | 6 | 6 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- T2D Participants (Panel B): Obese participants with T2D received once-weekly omarigliptin or placebo for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants - Omarigliptin | T2D Participants (Panel B) | T2D - Omarigliptin | T2D - Placebo | Total
Number analyzed (Participants) | 18 | 6 | 6 | 2 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (5.1) | 56.2 (7.6) | 55.4 (4.4) | 61.0 (8.5) | 54.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 3 | 1 | 20
  Male | 6 | 2 | 3 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Time Frame: Up to Day 36
Population: AEs were monitored in all obese healthy (Panel A) and Type 2 diabetes (T2D) (Panel B) participants who received omarigliptin 50 mg or placebo.
Measure: Number; unit: Participants
Groups:
- Healthy Omarigliptin: Obese healthy participants received once-weekly omarigliptin 50 mg for 4 weeks (Panel A).
- Healthy Placebo: Obese healthy participants received once-weekly placebo for 4 weeks (Panel A).
- T2D Omarigliptin: Obese participants with T2D received once-weekly omarigliptin 50 mg for 4 weeks (Panel B).
- T2D Placebo: Obese participants with T2D received once-weekly placebo for 4 weeks (Panel B).
Arm/Group | Healthy Omarigliptin | Healthy Placebo | T2D Omarigliptin | T2D Placebo
Number analyzed (Participants) | 18 | 6 | 6 | 2
Participants | 12 | 2 | 4 | 2

2. Primary Outcome: Number of Participants Withdrawing From Study Therapy Due to an AE
Time Frame: Up to Day 22
Population: AEs were monitored in all obese healthy (Panel A) and T2D (Panel B) participants who received omarigliptin 50 mg or placebo.
Measure: Number; unit: Participants
Arm/Group | Healthy Omarigliptin | Healthy Placebo | T2D Omarigliptin | T2D Placebo
Number analyzed (Participants) | 18 | 6 | 6 | 2
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percent Inhibition of Dipeptidyl Peptidase-4 (DPP-4) After Day 15
Description: Percent DPP-4 inhibition at 168 hours after the Day 15 dose (from baseline [pre-dose on Day 1]) was compared in healthy and T2D participants receiving omarigliptin or placebo.
Time Frame: 168 hours post-dose on Day 15
Population: Data from obese healthy participants (Panel A) and obese T2D participants (Panel B) 168 hours post-dose on Day 15 were pooled according to treatment. Predose data from Day 1 were missing from 2 participants.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent DPP-4 inhibition
Groups:
- Omarigliptin 50 mg: Obese healthy and T2D participants received once-weekly omarigliptin 50 mg for 4 weeks.
- Placebo: Obese healthy and T2D participants received once-weekly placebo for 4 weeks.
Arm/Group | Omarigliptin 50 mg | Placebo
Number analyzed (Participants) | 22 | 8
Percent DPP-4 inhibition | 91.92 [89.78 to 93.61] | 1.16 [-7.55 to 9.17]
Statistical Analysis 1: Comparison: Omarigliptin 50 mg vs Placebo; Test type: Superiority or Other; Difference in geometric means (GMs); Mean Difference (Final Values) = 90.76, 90% CI 2-sided [82.70 to 99.37]

4. Secondary Outcome: Percent Inhibition of DPP-4 After Day 22
Description: Percent DPP-4 inhibition at 168 hours after the Day 22 dose (from baseline [pre-dose on Day 1]) was compared in healthy and T2D participants receiving omarigliptin or placebo.
Time Frame: 168 hours post dose on Day 22
Population: No data from obese healthy participants (Panel A) were collected after pre-dose on Day 22. Therefore, data are presented only for obese T2D participants (Panel B) 168 hours post-dose on Day 22.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent DPP-4 inhibition
Arm/Group | Omarigliptin 50 mg | Placebo
Number analyzed (Participants) | 6 | 2
Percent DPP-4 inhibition | 89.62 [86.80 to 91.84] | -8.59 [-65.56 to 28.78]

5. Secondary Outcome: WAA Active Glucagon-like Peptide-1 (GLP-1) Concentration
Description: Weighted average augmentation (WAA) active GLP-1 concentration was based on the 0.25, 0.5, 1, 2, and 4 hour timepoints. WAA was calculated as area under the curve (AUC) for the 4-hr post-dose time period (AUC0-4 hrs); this AUC was then divided by the time interval of 4 hours to obtain WAA. Log scale data were then back-transformed to obtain LS means.
Time Frame: Through 4 hours post dose on Day 21
Population: Data from obese healthy participants (Panel A) and obese T2D participants (Panel B) 4 hours post dose on Day 21 were pooled according to treatment. All participants who received omarigliptin or placebo are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Omarigliptin 50 mg | Placebo
Number analyzed (Participants) | 24 | 8
pmol/L | 3.84 [3.38 to 4.36] | 2.0 [1.60 to 2.50]
Statistical Analysis 1: Comparison: Omarigliptin 50 mg vs Placebo; Test type: Superiority or Other; Ratio of geometric least-squares means = 1.92, 90% CI 2-sided [1.55 to 2.38] — GMR is ratio of active GLP-1 levels in omarigliptin:placebo groups

6. Secondary Outcome: WAA Total GLP-1 Concentration
Description: WAA total GLP-1 concentration was based on the 0.25, 0.5, 1, 2, and 4 hour timepoints. WAA was calculated as AUC0-4 hrs; this AUC was then divided by the time interval of 4 hours to obtain WAA. Log scale data were then back-transformed to obtain LS means.
Time Frame: Through 4 hours post dose on Day 21
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Omarigliptin 50 mg | Placebo
Number analyzed (Participants) | 24 | 8
pmol/L | 2.11 [1.82 to 2.44] | 2.31 [1.79 to 2.98]
Statistical Analysis 1: Comparison: Omarigliptin 50 mg vs Placebo; Test type: Superiority or Other; Ratio of geometric least-squares means = 0.91, 90% CI 2-sided [0.72 to 1.17] — GMR is ratio of total GLP-1 levels in omarigliptin:placebo groups

7. Secondary Outcome: Plasma Glucose Concentration
Description: Post-prandial glucose concentration is presented as a weighted average of the 0.25, 0.5, 1, 2, and 4 hour post-dose time points. Glucose concentration was calculated as area under the curve (AUC) for the 4-hr post-dose time period (AUC0-4 hrs); this AUC was then divided by the time interval of 4 hours to obtain weighted average glucose concentration. Log scale data were then back-transformed to obtain LS means.
Time Frame: Through 4 hours post dose on Day 21
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 50 mg | Placebo
Number analyzed (Participants) | 24 | 8
mg/dL | 8.34 [3.17 to 13.50] | 20.84 [11.90 to 29.78]

ADVERSE EVENTS:
Time Frame: Up to Day 36
Description: AEs were monitored up to 14 days after the final dose of study drug on Day 22.
Groups:
- Omarigliptin 50 mg Healthy (Panel A): Obese healthy participants received once-weekly omarigliptin 50 mg for 4 weeks.
- Placebo Healthy (Panel A): Obese healthy participants received once-weekly placebo for 4 weeks.
- Omarigliptin 50 mg T2D (Panel B): Obese T2D participants received once-weekly omarigliptin 50 mg for 4 weeks.
- Placebo T2D (Panel B): Obese T2D participants received once-weekly placebo for 4 weeks.
Arm/Group | Omarigliptin 50 mg Healthy (Panel A) | Placebo Healthy (Panel A) | Omarigliptin 50 mg T2D (Panel B) | Placebo T2D (Panel B)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 12/18 | 2/6 | 4/6 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 50 mg Healthy (Panel A) (N=18) | Placebo Healthy (Panel A) (N=6) | Omarigliptin 50 mg T2D (Panel B) (N=6) | Placebo T2D (Panel B) (N=2)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scintillating scotoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 1 (2) | 2 (5) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.